CLINICAL TRIAL: NCT04742192
Title: A Multicountry, Multicentre, Non-interventional, Prospective Study to Determine the Prevalence of EGFR Mutations in Patients With Early-stage, Surgically Resected, Non-squamous, Non-small Cell Lung Cancer
Brief Title: Non-interventional, Prospective Study to Determine Prevalence of EGFR Mutations in Non-small Cell Lung Cancer
Acronym: EARLY-EGFR
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D5161R00028
Record Dates: First submitted 2021-01-25; First posted 2021-02-08 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No

SUMMARY:
This prospective, multicountry, multicentre, non-interventional study plans to include patients who have undergone surgery for early-stage (IA to IIIB on the basis of pathologic criteria) non-squamous NSCLC up to 6 weeks prior to enrolment into the study.

The main objective of this study is to determine the prevalence of EGFRm in patients with surgically resected early-stage (IA to IIIB) non-squamous NSCLC as there are limited data on its prevalence in this patient population.

DETAILED DESCRIPTION:
This prospective, multicountry, multicentre, non-interventional study plans to include patients who have undergone surgery for early-stage (IA to IIIB on the basis of pathologic criteria) non-squamous NSCLC up to 6 weeks prior to enrolment into the study. Eligible patients should have availability of formalin-fixed paraffin-embedded (FFPE) specimen(s) to be primarily tested for EGFRm at validated local laboratories or a central laboratory. The informed consent will be obtained from the patients during their routine clinical care visit before data are collected from the medical records. The data on socio-demographics, tumour staging, histology, surgical management, and neoadjuvant therapies will be collected from available medical records at the treating facility by the investigator. If PD-L1 testing is conducted as part of routine clinical care, the available results will be recorded. Patients will be followed prospectively and follow-up will be considered as complete once EGFRm status of the patient's tumour sample is known and any planned adjuvant therapy has been recorded.

ELIGIBILITY:
Inclusion Criteria:

* Adult male or female patients ≥18 years old or 'adults' according to age of majority as defined by the local regulations
* Patient or next of kin/legal representative is willing and able to provide informed consent according to the local regulations, where applicable
* Patients with stage IA to IIIB (on the basis of pathologic criteria) NSCLC with adenocarcinoma, or mixed histology with an adenocarcinoma component who have undergone surgical resection of the tumour during the preceding 6 weeks
* Availability of FFPE tissue specimen suitable for EGFRm testing (either the primary diagnostic sample or the surgically resected tumour specimen)
* Availability of medical records at the participating site detailing the initial diagnosis, staging, and surgical management of NSCLC

Exclusion Criteria:

Patients who fulfil any of the following exclusion criteria will not be eligible for the study:

1. Histology of the tumour is considered not to be of primary lung in origin
2. Histology is pure squamous cell carcinoma, pure small cell carcinoma, or large cell carcinoma origin lacking any immunohistochemistry evidence of adenocarcinoma differentiation -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients who have stage IA to IIIB NSCLC with non-squamous histology and who have undergone surgical resection of tumour up to 6 weeks prior to enrolment
Sampling Method: Probability Sample
Enrollment: 601 (Actual)
Dates: Start 2021-03-04 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
Overall proportion of patients with EGFRm | 3 month
  Prevalence of EGFRm in patients with surgically resected early-stage (IA to IIIB on the basis of pathologic criteria) non-squamous NSCLC followed by Proportion of EGFRm by the following subgroup:
  o Histology (adenocarcinoma, bronchiole-alveolar, large cell carcinoma, mixed, other, unknown)
Proportion of EGFRm in Pathologic Stage | 3 Month
  Prevalence of EGFRm in patients with surgically resected early-stage (IA to IIIB on the basis of pathologic criteria) non-squamous NSCLC followed by Proportion of EGFRm by the following subgroup:
  o Pathologic stage (IA, IB, IIA, IIB, IIIA, IIIB with lymph node metastasis status [N0, N1, and N2])b

SECONDARY OUTCOMES:
Proportion of patients with the EGFRm types | 3 Month
  Proportion of patients with the following EGFRm types:
  * Exon19 deletions
  * Exon21 L858R
  * Exon20 T790M
  * Others (compound mutationsb, uncommon mutations [including G719X, L861Q, S768I, and 20 insertions])
Proportion of patients who were prescribed modalities | 3 Month
  Proportion of patients who were prescribed these modalities:
  * Only surgical resection
  * Surgical resection and radiotherapy
  * Surgical resection and systemic therapy (neoadjuvant and/or adjuvant)
  * Surgical resection, radiotherapy and systemic therapy (neoadjuvant and/or adjuvant)

OTHER OUTCOMES:
Proportion of patients with a tumour PD-L1 IHC test result | 3 Month
  Proportion of patients with PD-L1 positivity at various cut-points (<1%, ≥1%, ≥50%) grouped according to:
  * EGFRm
  * EGFR wild type

CONTACTS AND LOCATIONS:
Locations (31):
- Argentina (2):
  - Research Site, Rosario - Santa Fe, Argentina
  - Research Site, Buenos Aires
- Research Site, Santiago, Chile
- Colombia (2):
  - Research Site, Montería -Cordoba, Colombia
  - Research Site, Bogotá
- Research Site, San José, Costa Rica
- Research Site, Santo Domingo, Dominican Republic
- Egypt (3):
  - Research Site, Alexandria
  - Research Site, Cairo
  - Research Site, Tanta
- India (4):
  - Research Site, Kashmīr
  - Research Site, Kolkata
  - Research Site, Mumbai
  - Research Site, New Delhi
- Research Site, Kuwait City, Kuwait
- Mexico (3):
  - Research Site, Mexico City, Mexico City
  - Research Site, Guadalajara
  - Research Site, Monterrey
- Research Site, Lima, Peru
- Philippines (6):
  - Research Site, City of Taguig, Philippines
  - Research Site, Iliolo City, Philippines
  - Research Site, Cebu City
  - Research Site, Makati
  - Research Site, Manila
  - Research Site, Quezon City
- Research Site, Singapore, Singapore
- Thailand (2):
  - Research Site, Muang, Thailand
  - Research Site, Bangkok
- Research Site, Ankara, Turkey (Türkiye)
- Vietnam (2):
  - Research Site, Hanoi
  - Research Site, Ho Chi Minh City

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Batra U, Prabhash K, Noronha V, Deshpande R, Khurana S, Bhat GM, Mistry R, Agarwala V, Rajpurohit S, Poladia B, Sharma M, Banday SZ. Prevalence of EGFR Mutations in Patients With Resected Stage I to III Nonsquamous Non-Small Cell Lung Cancer: Results of India Cohort. JCO Glob Oncol. 2025 Jan;11:e2400353. doi: 10.1200/GO-24-00353. Epub 2025 Jan 7. PMID 39772802
- See also: Redacted CSR synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5161R00028&attachmentIdentifier=f8a9618e-fac2-4cf6-98db-e8ee04f49f59&fileName=EARLY-EGFR_Clinical_Study_Report_(CSR)_Synopsis_F.pdf&versionIdentifier=